CLINICAL TRIAL: NCT03863431
Title: The Influence of Overfeeding Different Macronutrients on Whole-body Insulin Sensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Carl Hulston, Senior Lecturer Nutrition and Metabolism, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R18-P222
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Insulin Resistance; Type 2 Diabetes; Glucose Metabolism Disorders; Metabolic Disease
Keywords: High-fat diets; High-carbohydrate diets; Glycaemic control
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Diet, High-Fat; Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat diet (Active Comparator): Participants will consume a diet rich in fat (approximately 65% of total energy) and low in carbohydrate for 14 days.
  Measurements will be made at 0, 7 and 14 days.
  Interventions: Other: High-fat diet
- High-carbohydrate diet (Active Comparator): Participants will consume a diet rich in carbohydrate (approximately 70% of total energy) and low in fat for 14 days.
  Measurements will be made at 0, 7 and 14 days.
  Interventions: Other: High-carbohydrate diet

INTERVENTIONS:
Other: High-fat diet — Participants will consume a high fat diet for 14 days with approximately 65% of energy from fat. The diet will also provide an energy excess, at 130% of energy requirements.
  Participants will be provided with all of their meals and snacks throughout the study.
  Arms: High-fat diet
Other: High-carbohydrate diet — Participants will consume a high fat diet for 14 days with approximately 70% of energy from carbohydrate. The diet will also provide an energy excess, at 130% of energy requirements.
  Participants will be provided with all of their meals and snacks throughout the study.
  Arms: High-carbohydrate diet

SUMMARY:
This study will investigate the effect of high-carbohydrate vs. high-fat overfeeding (130% of energy requirements) on whole body insulin sensitivity.

Following habitual diet, participants will be randomly allocated to either a high-carbohydrate or a high-fat diet intervention for 14-days. On days 0, 7 and 14 participants will undergo anthropometric and metabolic testing (primarily an oral glucose tolerance test [OGTT]).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* BMI = 18.5-29.9 kg/m2
* Male or female
* Physically active (> 3 x 30 min moderate exercise per week)
* Non-smoker (including the use of vaporisers and e-cigarettes)
* Healthy (determined by the School's standard health questionnaire)
* No cardiometabolic or inflammatory illness

Exclusion Criteria:

* Outside of age-range
* Outside BMI range
* Inactive (< 3 x 30 min moderate exercise per week)
* Smoker
* Taking medication
* History of cardiometabolic or inflammatory illness
* Vegetarian/ vegan (as the high-fat diet is based on animal fats)
* Other dietary restrictions which prevent consumption of the experimental diet
* Consumption of probiotics within last 3 months (these influence the gut microbiota)
* Participation in another clinical trial
* Those with known or suspected food intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Whole-body insulin sensitivity index | The change between pre-, during and post- dietary interventions: Assessed on days 0, 7 and 14
  Assessed by oral glucose tolerance test

SECONDARY OUTCOMES:
Body Mass Index | Day 0, Day 7, Day 14
  Calculated from height and weight
Fasting plasma glucose concentration | Day 0, Day 7, Day 14
  Measured in fasting plasma sample by spectrophotometric assay
Fasting serum insulin concentration | Day 0, Day 7, Day 14
  Measured in fasting serum sample by ELISA
Fasting plasma lipid profile (for example total and HDL cholesterol and TAG concentrations; all measured in mmol/L) | Day 0, Day 7, Day 14
  Measured in fasting plasma sample by spectrophotometric assay
Indirect calorimetry | Day 0, Day 7, Day 14
  Measured from expired gas samples
Subjective appetite ratings | Day 0, Day 7, Day 14
  Measured from visual analogue scale appetite questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Carl Hulston, PhD, Principal Investigator — Loughborough University
Locations (1):
- School of Sport, Exercise and Health Sciences, Loughborough, Leicestershire, United Kingdom